CLINICAL TRIAL: NCT01671423
Title: Use of a Single Dose of Oral Prednisone in the Treatment of Cellulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Principal Investigator, Scott Goldstein, DO, Attending Physician, Albert Einstein Healthcare Network
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HN 4372
Record Dates: First submitted 2012-08-14; First posted 2012-08-23 (Estimated); Results first posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-01

CONDITIONS: Cellulitis
Keywords: Cellulitis; Skin infection; Prednisone; Steroid; Anti-inflammatory
MeSH Terms: conditions — Cellulitis | interventions — Prednisone; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prednisone (Active Comparator): In addition to standard care for cellulitis, subject will receive a single 60 mg dose of Prednisone orally during their initial visit.
  Interventions: Drug: Prednisone
- Placebo (Placebo Comparator): In addition to standard care for cellulitis, subjects will receive a single placebo pill to take during their initial visit.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prednisone — See "Prednisone" arm description
  Other Names: Deltasone; Prednicot; Sterapred
  Arms: Prednisone
Drug: Placebo — See "Placebo" arm description
  Other Names: Sugar Pill; Inactive Drug; Control
  Arms: Placebo

SUMMARY:
Cellulitis is the medical term for an infection of the skin, with symptoms including redness, swelling, warmth, and pain. This group of symptoms is called inflammation, and is caused by the body's immune system responding to the infection. Standard care for cellulitis is using antibiotics to destroy the infection, but the inflammation can persist and cause a great deal of pain. The hypothesis of this study is that adding a single dose of an oral steroid (prednisone), which tempers the immune response, will reduce inflammation, reduce pain, and speed recovery. This hypothesis will be examined by recruiting a group of patients with cellulitis, and randomizing them to two sub-groups: one group will receive a dose of prednisone, while the other group will receive a placebo. Neither group will know what they received unless there is a problem. These subjects will be followed up at the 48 hour mark and the 7 day mark, and will have their results compared.

DETAILED DESCRIPTION:
This pilot study will be conducted in a prospective, double-blinded, placebo-controlled, randomized fashion using a convenience sample of 100 subjects who come to the ED with signs and symptoms of cellulitis. Initial medical assessment will be made by an attending/senior resident according with established clinical procedures, including the history, physical examination, and vital signs. If by clinical assessment the patients meet eligibility criteria, then they will be approached by a research associate for screening, informed consent process, enrollment in the study, and data collection.

After the subjects understand and sign the informed consent form, they will be randomized to either the placebo group or treatment group. The EMCP pharmacy will be in charge of the randomization process. Once randomized, a standard source document (see data management section and appendix C for details) will be filled with information given by the subjects and in their charts. While study medication is given (time zero), subjects will receive a Visual Analog Scale (VAS) to rate their pain upon initial presentation along with determination of size of the cellulitic area. This will be done by determining the longest axis of the cellulitic area and measuring it (in mm) from the most proximal/lateral end towards the most distal/medial end, excluding any lymphangitic spread. The most proximal and distal area of erythema will be outlined.

While the standard treatment of care for cellulitis will be circumscribed according to already established protocols, the class of antibiotics and pain control that patients receive will depend on their disposition:

If discharged:

1. Antibiotic prescriptions will be TMP/SMX 160/800 mg (Bactrim DS), 2 pills PO BID and Cephalexin 500 mg PO qid; if allergic, Clindamycin 300 mg PO QID.
2. Pain control: during stay in the ED subjects will receive, according to their allergic history and as long as the treating physician determines it is necessary to address the pain, two tablets of either Percocet 5/325 mg,Vicodin 5/500 mg (if allergic to Percocet), or Acetaminophen 500 mg as an only dose. Once discharged they will receive, according to their allergic history and the physician's clinical judgement, a prescription of 12 tablets of either Percocet 5/325 mg, Vicodin 5/500 mg (if allergic to Percocet), Tylenol #3 300/30 mg, or Acetaminophen 500 mg, one tablet PO q6 and PRN for pain. Pain medication must not include NSAIDs.

If admitted to observation unit: antibiotics will be IV Clindamycin 300 mg q6 hours; if allergic, IV Vancomycin 1 g q12 hours should be given. For pain control: Morphine 4 mg IV q4 hours and PRN pain; if allergic, Dilaudid 1 mg IV q4 hours and PRN if pain. Pain medication must not include NSAIDs. Once discharged, they will receive the same prescription as the discharged group of subjects.

In addition to the standard of care described and any additional medications deemed appropriate by the attending physician that do not represent a confounding factor to the study (NSAIDs, other antibiotics), subjects will also receive an additional pill which will be either prednisone 60 mg or placebo. If the treating physician feels it is in the best interest of the subject to break the protocol, the subject's participation in study procedures will end. Data that has already been collected will be kept, and may be analyzed separately. Once the subjects have received the study medications, they will follow their dispositions (either be discharged or be admitted in the observation's unit). To assure treatment compliance, the Research Associate will provide the subjects with antibiotics and pain medication treatment corresponding to the first 48 hours. After this landmark, the subjects will cover the rest of their treatment. Subjects will be instructed not to take any medication outside the prescription during the length of the study. If the subjects take NSAIDs during the first 48 hours, this could be considered a confounding factor. As such, subjects who take NSAIDs within the first 48 hours will have their participation in study procedures ended. Their already collected data will be kept and may be analyzed separately; however, if they take NSAIDs after the 48-hour visit their study participation will continue.

Subjects will be required to return to the ED after 48 hours and bring the remaining prescribed pain medications. They will meet a Research Associate for re-evaluation, which will be done by using a VAS, measuring the cellulitic area, and assessing the degree of usage of the prescribed pain medications. This second visit is not part of the standard of care so patients won't be required to receive a formal evaluation by an ED doctor nor register in triage. Financial compensation will be provided on completion of the 48 hour follow-up visit for all patients. A seventh (± one) day follow-up call will be done to assess pain severity, degree of symptomatic recovery and disappearance of the erythema, and need of additional medical assistance.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years
* Current episode of cellulitis

  1. Erythema greater than 5 centimeters in any dimension
  2. Pain, swelling, warmth, and tenderness in the area without elevated borders
* Dispositioned for discharge from the Emergency Department or Observation
* Able to consent

Exclusion Criteria:

* Steroid use in the past 2 weeks
* History of adrenal insufficiency
* Any infection treated with antibiotics in the past 2 weeks
* Allergy to:

  1. Steroids
  2. Acetaminophen
  3. Trimethoprim-Sulphamethoxazole (TMP/SMX), Cephalexin, and Clindamycin (must be allergic to all three for exclusion)
  4. Oxycodone and Hydrocodone (must be allergic to both for exclusion)
* If subject is going to the Observation unit, allergy to:

  1. Clindamycin and Vancomycin (must be allergic to both for exclusion)
  2. Morphine and Hydromorphone (must be allergic to both for exclusion)
* Suspicion or presence of abscess
* Suspicion or presence of deep vein thrombosis
* Suspicion or presence of severe sepsis, as defined by:

  1. Sepsis
  2. Hypotension (systolic pressure < 90 mmHg or reduction of 40 mmHg from baseline)
  3. Failure of single end organ
* Suspicion or presence of septic shock, as defined by:

  1. Severe sepsis
  2. Hypotension that is refractory to fluid management
  3. Failure or more than one end organ
* Crepitus
* Change in mentation
* Tachycardia greater than 120 beats per minute
* Fever greater than or equal to 39 degrees Celsius
* Hospital admission
* Under 18 years of age, or over 70 years of age
* Pregnancy or breast feeding
* Police custody or prisoner
* Cognitive impairment
* Inability to consent
* Nursing home residents

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Goldstein, DO, Principal Investigator — Albert Einstein Healthcare Network
Locations (1):
- Albert Einstein Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bergkvist PI, Sjobeck K. Antibiotic and prednisolone therapy of erysipelas: a randomized, double blind, placebo-controlled study. Scand J Infect Dis. 1997;29(4):377-82. doi: 10.3109/00365549709011834. PMID 9360253
- [Background] Kiderman A, Yaphe J, Bregman J, Zemel T, Furst AL. Adjuvant prednisone therapy in pharyngitis: a randomised controlled trial from general practice. Br J Gen Pract. 2005 Mar;55(512):218-21. PMID 15808038
- [Background] Qi D, Pulinilkunnil T, An D, Ghosh S, Abrahani A, Pospisilik JA, Brownsey R, Wambolt R, Allard M, Rodrigues B. Single-dose dexamethasone induces whole-body insulin resistance and alters both cardiac fatty acid and carbohydrate metabolism. Diabetes. 2004 Jul;53(7):1790-7. doi: 10.2337/diabetes.53.7.1790. PMID 15220203
- [Background] Todd KH, Funk KG, Funk JP, Bonacci R. Clinical significance of reported changes in pain severity. Ann Emerg Med. 1996 Apr;27(4):485-9. doi: 10.1016/s0196-0644(96)70238-x. PMID 8604867
- [Background] Yen MT, Yen KG. Effect of corticosteroids in the acute management of pediatric orbital cellulitis with subperiosteal abscess. Ophthalmic Plast Reconstr Surg. 2005 Sep;21(5):363-6; discussion 366-7. doi: 10.1097/01.iop.0000179973.44003.f7. PMID 16234700

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 42 participants agreed to participate in the study. Following completion of informed consent process, 1 participant withdrew of their own volition, 1 participant was excluded from analysis for taking NSAID within the first 48 hrs.
Period: Overall Study
Arm/Group | Prednisone | Placebo
Started | 20 | 20
Completed | 14 | 9
Not Completed | 6 | 11

BASELINE CHARACTERISTICS:
Population: Of the 40 subjects that were randomized, 25 subjects were analyzed; 14 received prednisone, 11 received placebo
Groups:
- Total: Total of all reporting groups
Arm/Group | Prednisone | Placebo | Total
Number analyzed (Participants) | 14 | 11 | 25
Age, Continuous [Mean (Full Range); unit: Years] — Population: Of the 40 subjects that were randomized, 25 subjects were analyzed; 14 received prednisone, 11 received placebo
  Years | 40 [21 to 58] | 40 [18 to 66] | 40 [18 to 66]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Of the 40 subjects that were randomized, 25 subjects were analyzed; 14 received prednisone, 11 received placebo
  Participants
    Female | 5 | 6 | 11
    Male | 9 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale(VAS) for Pain - Day 1 to 48 Hours
Description: The level of pain as measured by a Visual Analog Scale(VAS) measured once at day 1 and once during the 48th hour follow-up visit. Minimum value 0, maximum value 100mm, higher scores corresponds to more pain/worse outcomes.
Time Frame: Assessed once at day 1 and then once during the 48 hour follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 14 | 11
score on a scale
  VAS at Day 1 | 79.64 (14.89) | 56.45 (30.25)
  VAS at 48 hrs | 39.71 (34.5) | 25.91 (33.25)

2. Secondary Outcome: Amount of Pain Medication - Day 1 to 48 Hours
Description: Number of times the subject needed to use pain medication between day 1 and the 48 hour follow-up
Time Frame: Assessed once during the 48 hour follow-up
Population: Data is not available on all participants
Measure: Median (Full Range); unit: medications taken
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 14 | 11
medications taken | 7 [0 to 16] | 2 [0 to 12]

3. Secondary Outcome: Amount of Pain Medication - Day 1 to 7 Days
Description: Total amount of pain medication used between day 1 and the 7 day follow-up call.
Time Frame: Assessed once during the 7 day follow-up
Population: Data was not collected
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Amount of Pain Medication - 48 Hours to 7 Days
Description: Amount of pain medication the subject needed to use between the 48 hour follow-up and the 7 day follow-up.
Time Frame: Assessed at the 48 hour follow-up and at the 7 day follow-up
Population: Data was not collected
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants Requiring Additional Medical Assistance Post-Randomization
Description: Need for additional medical intervention to treat the current episode of cellulitis.
Time Frame: Assessed continuously from day 1 to the day 7 follow-up call
Population: Data was not collected
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Disposition Trend
Description: Disposition of the subject at the end of the initial visit on day 1; "Disposition Trend" refers to whether the subject was discharged to home or admitted to observation unit in the hospital. This Outcome Measure intends to assess improvement from baseline following intervention.
Time Frame: Assessed once during day 1
Population: Data is not available on all participants
Measure: Count of Participants; unit: Participants
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 14 | 11
Participants
  Discharged to Home | 12 | 8
  Data not available/not collected | 2 | 3

7. Secondary Outcome: Adverse Events (AE)
Description: Development of adverse events during study period such as: allergic reaction, development of severe sepsis or septic shock, crepitus, change in mentation, fever greater than or equal to 39 degrees Celsius, tachycardia (heart rate over 120 beats per minute)
Time Frame: Assessed continuously from day 1 to day 7 follow-up
Population: Data not collected on this outcome measure
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in Erythema Size - Day 1 to 48 Hours
Description: Change in erythema size - day 1 to 48 hours = (Mean erythema at Day 1) - (Mean erythema at 48 hrs) Erythema is measured in millimeters using the most proximal and distal area of the erythema. Higher values represent worse outcome.
Time Frame: Calculated once at 48 hrs
Population: Data not collected on this outcome measure
Arm/Group | Prednisone | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events collected upto 7 day follow up.
Arm/Group | Prednisone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
Small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes